CLINICAL TRIAL: NCT04385238
Title: Health and Wellbeing of Pregnant and Post-Partum Women During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Pregistry (Industry)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Other Study IDs: 0002
Record Dates: First submitted 2020-05-10; First posted 2020-05-12 (Actual); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: COVID-19; Pregnancy Complications; Mental Health Wellness 1; Anxiety; Depression; Ptsd; Coronavirus
MeSH Terms: conditions — COVID-19; Pregnancy Complications; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Women: Pregnant women who are 18 years of age or older.
  Interventions: Other: This is an online survey with no intervention.
- Post-partum women: Women who gave birth within the last 6 months who are 18 years of age or older.
  Interventions: Other: This is an online survey with no intervention.

INTERVENTIONS:
Other: This is an online survey with no intervention. — As this is an online survey about health and wellbeing, there is no intervention.

SUMMARY:
The purpose of this study is to assess the health and wellbeing of pregnant and recently pregnant women during the COVID-19 pandemic using an online survey.

DETAILED DESCRIPTION:
Millions of women will give birth during the pandemic of Coronavirus Disease 2019 (COVID-19) caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The consequences of COVID-19 for pregnant women and their offspring are unknown. This lack of information leads to anxiety among pregnant women, women who are considering getting pregnant, and their families. It is therefore important to assess the wellbeing and mental health of women during the COVID-19 pandemic.

The international nature of the online survey will allow the evaluation of how living during the COVID-19 pandemic affects pregnant and recently pregnant women at a global level, including the evaluation of potential cultural and geographic differences.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women or women who have been pregnant within the last 6 months
* Able to give electronic informed consent

Exclusion Criteria:

* <18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Persons assigned gender female at birth.
Study Population: Pregnant women or women who have been pregnant in the last 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 6894 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karestan Koenen, PhD, Principal Investigator — Department of Epidemiology, Harvard T.H. Chan School of Public Health; Sonia Hernandez-Diaz, MD, DrPh, Study Director — Department of Epidemiology, Harvard T.H. Chan School of Public Health; Diego Wyszynski, MD, MHS, PhD, Study Director — Pregistry
Locations (1):
- Pregistry, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Survey Health and Wellbeing of Pregnant and Post-Partum Women During the COVID-19 Pandemic — https://survey.pregistry.com/
- See also: International Registry of Coronavirus Exposure in Pregnancy (IRCEP) — https://corona.pregistry.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregnant Women | Post-partum Women
Started | 5712 | 1182
Completed | 5712 | 1182
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnant Women | Post-partum Women | Total
Number analyzed (Participants) | 5712 | 1182 | 6894
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (4.1) | 31.7 (4.9) | 31.3 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5712 | 1182 | 6894
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1288 | 131 | 1419
  Not Hispanic or Latino | 4424 | 1051 | 5475
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptoms of Post-traumatic Stress Disorder
Description: Post-traumatic Stress Disorder (PTSD) Symptoms will be assessed by the Impact of Events Scale-6. This scale includes a total of six items: two items from each of the three subscales of the measure, namely intrusion, hyperarousal and avoidance. Participants will be asked to report their PTSD symptoms in the past 7 days on a Likert Scale ranging from 0 (not at all) to 4 (extremely).
Time Frame: Anytime during pregnancy or within 6 months after given birth.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women | Post-partum Women
Number analyzed (Participants) | 5712 | 1182
Participants | 1028 | 532

2. Primary Outcome: Number of Participants With Symptoms of Anxiety and Depression
Description: Symptoms of anxiety and depression will be measured by the Patient Health Questionnaire-4 (PHQ-4) which combines two ultrabrief screeners: the PHQ-2 and the Generalised Anxiety Disorder Scale. Participants will be asked to report their symptoms of depression and anxiety in the past 2 weeks on a Likert Scale from 0 (not at all) to 3 (nearly every day) for a maximum score of 12.
Time Frame: Anytime during pregnancy or within 6 months after given birth.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women | Post-partum Women
Number analyzed (Participants) | 5712 | 1182
Participants | 1200 | 438

ADVERSE EVENTS:
Time Frame: This is a cross-sectional observational survey and, therefore, adverse event data were not collected.
Description: This is a cross-sectional observational survey and, therefore, adverse event data were not collected.
Groups:
- Pregnant Women: Pregnant women who are 18 years of age or older.
  This is an online survey with no intervention: As this is an online survey about health and wellbeing, there is no intervention and no assessment of adverse events.
- Post-partum Women: Women who gave birth within the last 6 months who are 18 years of age or older.
  This is an online survey with no intervention: As this is an online survey about health and wellbeing, there is no intervention and no assessment of adverse events.
Arm/Group | Pregnant Women | Post-partum Women
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT04385238/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT04385238/SAP_001.pdf